CLINICAL TRIAL: NCT01814098
Title: Escitalopram in the Long-term Treatment of Major Depressive Disorder With Associated Anxiety Symptom
Brief Title: An Efficacy and Safety Study of Escitalopram Long-Term Treatment in Major Depressive Disorder With Associated Anxiety Symptoms
Acronym: Lexapro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016381; ESCITALDEP4002
Record Dates: First submitted 2013-03-14; First posted 2013-03-19 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Escitalopram; Lexapro
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Escitalopram (Experimental): Escitalopram tablets will be administered orally at 10 milligram per day (mg/day). The dose may be increased to maximum of 20 mg/day depending on Investigators discretion for 24 weeks
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram tablets will be administered orally at 10 milligram per day (mg/day). The dose may be increased to maximum of 20 mg/day depending on Investigators discretion for 24 weeks
  Other Names: Lexapro

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of long term escitalopram treatment in participants with Major Depressive Disorder (MDD) with associated anxiety symptoms.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single arm, prospective (study following participants forward in time), post-marketing, multi-center (when more than one hospital or medical school team work on a medical research study) study to evaluate the efficacy and safety of escitalopram in participants with MDD with associated anxiety symptoms. The duration of the study will be 24 weeks at a starting dose of escitalopram 10 milligram per day (mg/day). The dose will be flexibly adjusted (maximum 20 mg/day) after 2 weeks of treatment depending on Investigator's discretion. The study will consist of 9 visits: Baseline, Week 1, 2, 4, 8, 12, 16, 20 and 24. Assessments of efficacy and safety will be performed at each visit. The primary efficacy evaluation will be done by Montgomery-Asbery Depression Rating Scale (MADRS) and Hamilton Anxiety Scale(HAM-A). Participant's safety will also be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be willing and able to give written informed consent
* Participant currently suffering from Major Depressive Disorder (MDD) with anxious symptoms including participant with first MDD episode, and relapsed participant with new episode
* Participant with minimum score at baseline of 22 on the Montgomery-Asbery Depression Rating Scale (MADRS) and minimum score at baseline of 14 on Hamilton Anxiety Rating (HAM-A) scales
* Female participant must be surgically sterile, or practicing an effective method of birth control before entry and throughout the study

Exclusion Criteria:

Participant who has continuously taken psychoactive substances, antidepressants, anxiolytics, monoamine oxidase inhibitors (MAOIs), psychoactive herbal remedies, lithium, electroconvulsive therapy (ECT) carbamazepine in the past 2 weeks before the baseline visit - Participants with MDD, requiring treatment systematically within past 2 months from baseline - Participants who has contraindication to escitalopram - Participant has primary or comorbid diagnoses of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations [imagining things], and withdrawal into the self), schizoaffective disorder (a mixed psychiatric disorder relating to a complex psychotic state that has features of both schizophrenia and a mood disorder such as bipolar disorder), bipolar disorder, or dementia (mental decline) - Participant who has a significant risk of suicide on clinical assessment or has made a serious suicide attempt within the past 6-month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2009-07-07 (Actual); Primary Completion 2011-05-31 (Actual); Study Completion 2011-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Remission According to Montgomery-Asbery Depression Rating Scale (MADRS) and Hamilton Anxiety Scale (HAM-A) | Week 24
  Remission is defined as MADRS total score =<10 and HAM-A score =<7. MADRS measures depression severity and detects changes due to antidepressant treatment. It consists of 10 items, each scoring from 0 (not present) to 6 (severe). Total score= 0-60. Higher scores indicate more severe condition. HAM-A is 14-item scale measuring anxiety in individuals. Each question reflects a symptom of anxiety (physical and mental symptoms). The answers range from 0 (complete lack of symptom) to 4 (very severe show of anxiety with that symptom). Total score= 0-56. Higher scores indicate a more severe condition.

SECONDARY OUTCOMES:
Percentage of Participants Showing Response | Week 24
  Response is defined as having more than or equal to 50 percent decrease from baseline of MADRS total score. The MADRS is a scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change From Baseline in MADRS Total Score at Week 24 | Baseline and Week 24
  The MADRS is a scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change From Baseline of Single Rating Item in MADRS Total Score at Week 24 | Baseline and Week 24
  The MADRS is a scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Change From Baseline in Hamilton Depression Rating Scale (HAMD)-17 Score at Week 24 | Baseline and Week 24
  The depressive symptoms will be assessed using the 17-item HAMD scale, which provides a total score (0-52) (sum of the scores of all 17 items ). For total score of each item, higher score indicates severity of depressive symptom.
Change From Baseline in Hamilton Anxiety Scale (HAM-A) Score at Week 24 | Baseline and Week 24
  The HAM-A is a 14-item scale designed to measure anxiety in individuals,which provide a total score of 0-56. Higher scores indicate a more severe condition. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. The answers range from 0 which signifies a complete lack of that symptom to 4, which indicates a very severe show of anxiety with that symptom.
Change From Baseline of Single Rating Item in HAM-A at Week 24 | Baseline and Week 24
  The HAM-A is a 14-item scale designed to measure anxiety in individuals,which provide a total score of 0-56. Higher scores indicate a more severe condition. Each question reflects a symptom of anxiety and physical as well as mental symptoms are represented. The answers range from 0 which signifies a complete lack of that symptom to 4, which indicates a very severe show of anxiety with that symptom.
Change From Baseline in Clinical Global Impression Score (CGI-S) at Week 24 | Baseline and Week 24
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.
Change From Baseline in Short Form-12 (SF-12) Score at Week 24 | Baseline and Week 24
  The SF-12 consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health Each item is scored into on a 0-100 range. All items are scored so that a high score defines a more favorable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.
Locations (10):
- China (10):
  - Beijng
  - Changsha
  - Hangzhou
  - Nanjing
  - Shanghai
  - Shenyang
  - Shijiazhuang
  - Tianjin
  - Wenzhou
  - Wuhan

REFERENCES:
- See also: Escitalopram in the Long-term Treatment of Major Depressive Disorder With Associated Anxiety Symptom — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2348&filename=CR016381_CSR.pdf